CLINICAL TRIAL: NCT04193384
Title: Analysis of Weight Regain Rate and Predictive Factors in Patients Submitted to Bariatric Surgery.
Brief Title: Predictive Factors of Regain in Bariatric Patients Without Outpatients Care Regular.
Acronym: Obesity
Status: Completed | Type: Observational
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Luiz Guilherme Kraemer-Aguiar, MD, Professor, Rio de Janeiro State University
Other Study IDs: BAREG
Record Dates: First submitted 2019-12-04; First posted 2019-12-10 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Obesity; Bariatric Surgery
Keywords: Obesity; Bariatric Surgery; Weight Gain; Predictive Factors
MeSH Terms: conditions — Obesity; Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1≤ (G1≤): Group 1≤ (G1≤) - patients that performed bariatric surgery for ≤ 1 year
- Group 1> (G1>): Group 1> (G1>) - patients that performed bariatric surgery for > 1 year

SUMMARY:
The bariatric surgery is recommended for treatment of patients with severe obesity, resulting in greater weight loss and improvement of cardiovascular and metabolic comorbidities. However, weight regain is observed in patients after surgery, leading to health adverse outcomes. The purpose of this study is to identify the rate of weight regain and predictive factors of regain in bariatric patients without outpatients care regular.

DETAILED DESCRIPTION:
Post-bariatric patients without care by health professional will be recruited. Patients will be divided, initially, in two groups by time after surgical procedure, as follows: Group 1≤ (G1≤) - patients that performed bariatric surgery for ≤ 1 year and Group 1> (G1>) - patients that performed bariatric surgery for > 1 year. Patients will be seen in a medical set for the first time at the Policlínica Piquet Carneiro (PPC) for outpatients care, which will consist of anamnesis and physical examination, obtaining demographic, socioeconomic data, medications and clinical history. The TxR will be calculated by [TxR = (current weight - minimum weight reported) x 100 / (weight preoperatively reported - minimum weight related)] and information on predictive variables for weight regain will be obtained by Alcohol Use Disorders Identification Test (AUDIT), Beck Depression Inventory (BDI), International Physical Activity Questionnaire (IPAQ), ActiGraph GT3X + accelerometer, 36-Item Short-Form Health Survey (SF-36), Eating Disorder Examination-Questionnaire (EDE-Q) and Repetitive eating questionnaire (REP(EAT) Q). The inclusion period of new patients in the PPC Obesity Clinic will be one year.

ELIGIBILITY:
Inclusion Criteria:

- Bariatric patients without regular medical follow-up

Exclusion Criteria:

* Pregnancy
* Bariatric patients under one year of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Post-bariatric patients without care by health professional with more than one year of surgery.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Analysis of the association between weight regain and alcohol abuse disorder | through study completion, an average of 1 year
  Analysis of the association between weight regain (weight in kg) and Alcohol abuse (avaliated by Alcohol Use Disorders Identification Test) in the first clinical evaluation
Analysis of the association between weight regain and general psychopathology | through study completion, an average of 1 year
  Analysis of the association between weight regain (weight in kg) and general psychopathology (avaliated by Beck Depression Inventory) in the first clinical evaluation
Analysis of the association between weight regain and physical activity level | through study completion, an average of 1 year
  Analysis of the association between weight regain (weight in kg) and physical activity (avaliated by International Physical Activity Questionnaire and the ActiGraph accelerometer) in the first clinical evaluation
Analysis of the association between weight regain and quality of life indicators | through study completion, an average of 1 year
  Analysis of the association between weight regain (weight in kg) and quality of life (avaliated by the 36-Item Short-Form Health Survey Questionnaire) in the first clinical evaluation
Analysis of the association between weight regain and eating Disorder | through study completion, an average of 1 year
  Analysis of the association between weight regain (weight in kg) and eating disorder (avaliated by Eating Disorder Examination-Questionnaire and Repetitive eating questionnaire) in the first clinical evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory for Clinical and Experimental Research on Vascular Biology, Rio de Janeiro State University, Rio de Janeiro, Rio de Janeiro, Brazil, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopes KG, Dos Santos GP, Romagna EC, Mattos DMF, Braga TG, Cunha CB, Maranhao PA, Kraemer-Aguiar LG. Changes in appetite, taste, smell, and food aversion in post-bariatric patients and their relations with surgery time, weight loss and regain. Eat Weight Disord. 2022 Jun;27(5):1679-1686. doi: 10.1007/s40519-021-01304-3. Epub 2021 Sep 23. PMID 34554440